CLINICAL TRIAL: NCT04965831
Title: Furmonertinib Mesylate as Perioperation Therapy in Stage IIIA-IIIB (N1-N2) Resectable, EGFR Sensitizing Mutation Positive Lung Adenocarcinoma Patients: A Phase II, Single-arm, Open-label Clinical Study (FRONT)
Brief Title: Furmonertinib as Perioperation Therapy in Stage IIIA-IIIB (N1-N2) Resectable EGFR Mutated Lung Adenocarcinoma (FRONT)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AST-PMR2003
Record Dates: First submitted 2021-06-27; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (Experimental): Furmonertinib as perioperation therapy
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 80mg/d as neoadjuvant therapy for 8 weeks before surgery, then as adjuvant therapy for 3 years after surgery.
  Other Names: AST2818

SUMMARY:
This is a phase II study aimed to assess the efficacy and safety of furmonertinib, a third generation EGFR TKI, as perioperation therapy in stage IIIA-IIIB (N1-N2) resectable NSCLC patients.

DETAILED DESCRIPTION:
Please refer to detailed description in the following context.

ELIGIBILITY:
Inclusion Criteria:

* The written informed consent of the patients has been obtained before any examination, sampling and analysis related to the study.
* Primary lung adenocarcinoma diagnosed histologically/cytologically.
* Stages IIIA-IIIB (N1-N2) according to the AJCC 8th edition lung cancer stage and plan to receive radical excision judged by investigators.
* EGFR mutation positive (19Del or L858R, with or without T790M)
* The presence of at least one measurable lesion and suitable for accurate repeated measurements.
* ECOG performance status 0-1.
* For premenopausal women with fertility, the result of serum or urine pregnancy test should be negative within 7 days before the first dose.

Exclusion Criteria:

* Squamous cell carcinoma, and tumors with neuroendocrine components such as large cell carcinoma, or small cell carcinoma.
* Patients with EGFR exon 20 insertion mutation.
* Exposure to other antitumor therapies prior to enrolment.
* Major surgery was performed in the four weeks prior to the first dosing of the study drug.
* Pregnant or lactating female patients.
* Use of CYP3A4 strong depressant within 7 days or CYP3A4 strong inducer within 21 days prior to initial administration.
* Have a history of or present complications with other malignancies.
* Patients with severe or uncontrolled systemic disease requiring treatment were not considered suitable for the study.
* ECG QT interval prolongation or associated risk.
* A history of interstitial pneumonia or related risk.
* Inadequate bone marrow or organ reserve.
* Other circumstances that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 8 weeks following the first dose of study drug
  Proportion of patients whose tumors were assessed as complete response(CR) or partial response(PR) according to RECIST 1.1

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Approximately 8 weeks following the first dose of study drug
  Proportion of patients whose tumors were assessed as CR, PR or stable disease (SD) according to RECIST 1.1
Progression free survival (PFS) | Approximately 3 years following the first dose of study drug
  The time from the first does of the study drugs to the progression of the disease or death for any reason.
Disease free survival (DFS) | Approximately 3 years following the first dose of study drug
  The time from the end of surgery to the progression of the disease or death for any reason.
Adverse Events (AEs) | From the start of study drug to 28 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0

OTHER OUTCOMES:
Circulating tumor DNA clearance rate | Approximately 8 weeks following the first dose of study drug
  The proportion of patients with circulating tumor DNA clearance after neoadjuvant therapy
Minimal residual disease rate | Approximately 12 weeks following the first dose of study drug
  The proportion of patients with minimal residual disease defined as detectable ctDNA with a variant allele fraction of at least 0.1% in plasma after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan is not to be shared according to the policy.